CLINICAL TRIAL: NCT03628794
Title: Pilot Testing the Digital Supportive Care Awareness & Navigation (D-SCAN) Application
Brief Title: Digital Supportive Care Awareness & Navigation
Acronym: D-SCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00092123
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-04

CONDITIONS: Supportive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Subjects in the intervention group will receive the D-SCAN mobile application
  Interventions: Device: D-SCAN
- Control (Other): Subjects randomized into the control group will receive standard of care which includes the routine provision of information about supportive care services by nurses and other staff in the DCI clinics, as part of the standard nurse-driven distress screening and management process
  Interventions: Device: D-SCAN

INTERVENTIONS:
Device: D-SCAN — Subjects will receive a digital patient navigator service in the form of a mobile application ("app"), which has been designed at Duke, with feedback from Duke Cancer Institute (DCI) patients, caregivers and clinicians. Its purpose is to facilitate awareness of available Cancer Patient Support Program (CPSP) services at Duke, and to also help patients recognize their unmet symptom management needs. Subjects receiving the D-SCAN mobile app will also complete a survey every week within the app. The first 15 patients and 5 caregivers randomized into the intervention arm (those receiving the app) will also be asked to participate in a qualitative interview assessment at week 12, +/- 3 weeks

SUMMARY:
To pilot test the feasibility, usability, and preliminary efficacy of the D-SCAN mobile application in cancer patients and caregivers at Duke.

DETAILED DESCRIPTION:
D-SCAN, a digital patient navigator service in the form of a mobile application ("app"), has been designed at Duke, with feedback from Duke Cancer Institute (DCI) patients, caregivers and clinicians (screenshots in Appendix A).3 Its purpose is to facilitate awareness of available Cancer Patient Support Program (CPSP) services at Duke, and to also help patients recognize their unmet symptom management needs by answering questions from the Edmonton Symptom Assessment Scale (ESAS). This novel electronic system helps to connect patients and their loved ones with existing resources tailored to their unique situations, ensuring that no supportive care needs go unaddressed, thus improving patients' lives and their cancer care.

This protocol aims to assess the feasibility, usability, and preliminary efficacy of the D-SCAN mobile application. The app data, along with quantitative and qualitative feedback obtained during the pilot, will inform future development and design of a subsequent efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least age 18
* Patients who have the capacity to give consent
* Patients with advanced cancer who have initiated treatment at the DCI in the last 12 weeks
* Caregivers over the age of 18 caring for either enrolled or not enrolled patients with advanced cancer who have initiated treatment at the DCI in the last 12 weeks

Exclusion Criteria:

* Patients who are too ill to participate (per clinician discretion)
* Patients not able to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Number of enrolled patients complete at least 3 of the 12 symptom surveys over the study duration | 12 weeks
Number of patients who complete the exit survey | 12 weeks
Number of patients who return the phone | 12 weeks

SECONDARY OUTCOMES:
Frequency of use | 12 weeks
Duration of use | 12 weeks
Session Length | 12 weeks
Number of content views | 12 weeks
Number of actions taken | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Merz A, Mohamed A, Corbett C, Herring K, Hildenbrand J, Locke SC, Patierno S, Troy J, Wolf S, Zafar SY, Chilcott J, Higgins A, Manassei H, McCoy C, Buckingham TL, LeBlanc TW. A single-site pilot feasibility randomized trial of a supportive care mobile application intervention for patients with advanced cancer and caregivers. Support Care Cancer. 2022 Oct;30(10):7853-7861. doi: 10.1007/s00520-022-07224-x. Epub 2022 Jun 20. PMID 35718794